CLINICAL TRIAL: NCT04408937
Title: A Randomized, Investigator and Subject Blinded, Multicenter, Parallel-arm Study to Determine the Safety and Tolerability of Tropifexor.
Brief Title: The Purpose of This Study is to Investigate Safety and Tolerability of Tropifexor.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLJN452A2113
Record Dates: First submitted 2020-05-28; First posted 2020-05-29 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Liver Disease
Keywords: tropifexor; FXR agonist
MeSH Terms: conditions — Liver Diseases | interventions — tropifexor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- tropifexor AM 200 micrograms and Placebo (PM) (Experimental): Tropifexor 200 μg (AM) and Placebo (PM) once daily each
  Interventions: Drug: triopifexor; Drug: Placebo
- tropifexor PM 200 micrograms and Placebo (AM) (Experimental): Tropifexor 200 μg (PM) and Placebo (AM) once daily each
  Interventions: Drug: triopifexor; Drug: Placebo

INTERVENTIONS:
Drug: triopifexor — Tropifexor as a dry blend in hard gelatin capsules for oral administration
  Other Names: LJN452
Drug: Placebo — Placebo capsules for oral administration

SUMMARY:
The purpose of this study is to determine whether dosing tropifexor is safe and tolerable.

DETAILED DESCRIPTION:
This was a randomized, subject and investigator blinded, multicenter, parallel-arm study to assess the safety and tolerability of tropifexor dosed in the evening as compared to dosing in the morning in subjects with non-alcoholic steatohepatitis (NASH). Subjects whose eligibility was confirmed were randomized with stratification by domicile status at Day 1 of the treatment period into tropifexor (200 μg) AM dose group (hereafter referred to as AM dose group) or tropifexor (200 μg) PM dose group (hereafter referred to as PM dose group) in a 1:1 ratio. Subjects in the AM dose group took tropifexor in the morning and placebo in the evening while subjects in the PM dose group took placebo in the morning and tropifexor in the evening for 4 weeks in a blinded manner.

ELIGIBILITY:
Inclusion Criteria:

-Presence of Liver Disease

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations.
* Subjects taking the following medicines UNLESS on a stable dose (within 25% of baseline dose) for at least 3 months before randomization:

Type 1 diabetes and Uncontrolled Type 2 diabetes defined as Glycated hemoglobin (HbAlc) ≥ 9.5% at screening

-Calculated estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73m2 (using the Modification of diet in renal disease (MDRD) formula) Subjects with contraindications to Magnetic resonance imaging (MRI) imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fasting circulating LDL-C levels after 2 weeks of tropifexor treatment | week 2

SECONDARY OUTCOMES:
Change in fasting circulating High density lipoprotein cholesterol (HDL-C) and low density lipoprotein cholesterol (LDL-C) levels over 4 weeks of treatment | week 4
Change in ALT, AST and GGT over 4 weeks of treatment | week 4
PK parameters include but not limited to Cmax (ng/ml) will be assessed in the domiciled patients | week 4
PK parameters include but not limited to area under the curve (AUC) will be assessed in the domiciled patients | 4 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Novartis Investigative Site, Madison, Alabama
  - Novartis Investigative Site, Coronado, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, South Bend, Indiana
  - Novartis Investigative Site, Morehead City, North Carolina
  - Novartis Investigative Site, Hermitage, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=975
- See also: Results for CLJN452A2113 can be found on the Novartis Clinical Trial Results Website. — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17871